CLINICAL TRIAL: NCT05462067
Title: Visual Performance of Patients With Either Bilateral Implantation of the ZEISS AT LARA or the ZEISS AT LARA in One Eye and ZEISS AT LISA Tri in the Other (Presbyopia IOL Concept Evaluation).
Brief Title: Combined EDOF / Trifocal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GPAS-LARALISA-2018-01
Record Dates: First submitted 2022-07-04; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Binocular EDOF IOL (Active Comparator): Binocular EDOF IOL for treatment of cataract
  Interventions: Device: AT LARA IOL
- Combined Edof and Trifocal IOL (Experimental): Combined EDOF and Trifocal IOL - EDOF in the distance dominant eye / Trifocal in the non-dominant eye
  Interventions: Device: AT LARA IOL; Device: AT LISA Tri IOL

INTERVENTIONS:
Device: AT LARA IOL — EDOF IOL for treatment of cataract
Device: AT LISA Tri IOL — Trifocal IOL for treatment of cataract
  Arms: Combined Edof and Trifocal IOL

SUMMARY:
The purpose of this study is to obtain postoperative visual performance data of patients with bilateral implantation of the AT LARA IOL or the AT LARA implanted in the dominant eye and AT LISA tri implanted in the other eye. Dependence on spectacles, the occurrence of photic phenomena and patient and surgeon satisfaction with the patient's visual performance will be documented. Furthermore, the refraction data will be used to optimize the IOL constants for IOL power calculations.

DETAILED DESCRIPTION:
An extended depth of field can enable patients to do most everyday tasks without glasses. Compared to MIOLs, side effects such as glare and halo perception are expected to be less frequent and with lower intensity. This study is designed to assess visual performance and satisfaction in patients who underwent bilateral AT LARA IOL implantation or a mixed implantation of AT LARA in the dominant eye and AT LISA tri in the non-dominant eye. All patients will be offered enrolment after successful implantation in both eyes. Therefore, the preoperative and surgical data are recorded retrospectively, the follow-up examinations will be documented prospectively. This approach is justified and does not cause bias, as the purpose of this study is to investigate the performance of the IOL after successful implantation and uncomplicated surgery.

In this retrospective/prospective, non-randomized study, subjects will receive either binocular implantation of AT LARA/AT LARA toric or AT LARA/AT LARA toric in the distance dominant eye and AT LISA tri/AT LISA tri toric in the non-dominant eye. The main outcome parameter is best corrected visual acuity (CDVA). Secondary outcome parameters are: preferred near and intermediate distance, UDVA, DCIVA (Salzburg Reading desk in preferred distance), DCNVA (Salzburg Reading Desk in preferred near distance), distance corrected intermediate and near visual acuity with different contrast settings (Salzburg Reading Desk), manifest refraction, monocular and binocular defocus curve analysis, dysphotopsia simulation (Halo & Glare Simulator), subjective patient satisfaction (MacAlinden) questionnaire.

Patients have different demands for intermediate and near vision as well as distances needed for daily routine. Comparing both groups indicates there is individual lens fitting for patients depending on their own needs. Subjects are to be evaluated 2-4 months and 5-8 months after implantation of either configuration.

ELIGIBILITY:
Inclusion Criteria:

* Patients bilaterally implanted with the AT LARA IOL or the AT LARA and AT LISA tri IOLs or their toric versions
* Age 18 and older
* Uncomplicated implantation of study IOLs
* No visual acuity limiting pathologies
* Clear intraocular media
* Availability, willingness and sufficient cognitive awareness to comply with examination procedures
* Written informed consent for participation in the study and data protection

Exclusion Criteria:

* Visual potential of less than 0.63 (decimal) in each eye due to ocular pathologies, e.g. retinal disorders
* Postoperative CDVA >0.2 log MAR
* Visual field loss which has impact on visual acuity
* Use of systemic or ocular medication that might affect vision
* Acute or chronic disease, illness, ocular trauma or surgery that would confound results (e.g. macular degeneration, cystoid macular edema, proliferative diabetic retinopathy, etc.)
* Patients with amblyopia, strabismus, forme fruste keratoconus or keratoconus
* Capsular or zonular abnormalities that have affected postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome)
* Pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils, or pupils that do not dilate at least 3.5 mm under mesopic/scotopic conditions)
* Patient participates in other clinical trial (former participation is no exclusion criterion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Change in preoperative and postoperative binocular Corrected Distance Visual Acuity (CDVA) | Pre-op, 2-4 Months, & 5-8 Months
  The uncorrected and best corrected distance visual acuity is determined with standard reading charts at a distance of 4 or 5 m; logMar visual acuity is recorded.
  Near visual acuity (40 cm) and intermediate visual acuity (67 cm) are documented using suitable visual acuity charts for the respective distance or converted using conversion tables. The logMar visual acuity is recorded.
  Uncorrected visual acuity will be scored for distance, intermediate and near vision:
  * logMAR 0.0 or better = 5
  * logMar 0.1 = 4
  * logMar 0.2 = 3
  * logMar 0.3 = 2
  * logMAR worse than 0.3 = 1 Scores for the individual distances will be added to a total score.

SECONDARY OUTCOMES:
Postoperative uncorrected monocular and binocular distance visual acuity | 2-4 Months, & 5-8 Months
  The uncorrected and best corrected distance visual acuity is determined with standard reading charts at a distance of 4 or 5 m; logMar visual acuity is recorded.
  Near visual acuity (40 cm) and intermediate visual acuity (67 cm) are documented using suitable visual acuity charts for the respective distance or converted using conversion tables. The logMar visual acuity is recorded.
  Uncorrected visual acuity will be scored for distance, intermediate and near vision:
  * logMAR 0.0 or better = 5
  * logMar 0.1 = 4
  * logMar 0.2 = 3
  * logMar 0.3 = 2
  * logMAR worse than 0.3 = 1 Scores for the individual distances will be added to a total score.
Postoperative uncorrected and distance-corrected binocular near visual acuity | 2-4 Months, & 5-8 Months
  The uncorrected and best corrected distance visual acuity is determined with standard reading charts at a distance of 4 or 5 m; logMar visual acuity is recorded.
  Near visual acuity (40 cm) and intermediate visual acuity (67 cm) are documented using suitable visual acuity charts for the respective distance or converted using conversion tables. The logMar visual acuity is recorded.
  Uncorrected visual acuity will be scored for distance, intermediate and near vision:
  * logMAR 0.0 or better = 5
  * logMar 0.1 = 4
  * logMar 0.2 = 3
  * logMar 0.3 = 2
  * logMAR worse than 0.3 = 1 Scores for the individual distances will be added to a total score.
Postoperative uncorrected and distance-corrected binocular intermediate visual acuity | 2-4 Months, & 5-8 Months
  The uncorrected and best corrected distance visual acuity is determined with standard reading charts at a distance of 4 or 5 m; logMar visual acuity is recorded.
  Near visual acuity (40 cm) and intermediate visual acuity (67 cm) are documented using suitable visual acuity charts for the respective distance or converted using conversion tables. The logMar visual acuity is recorded.
  Uncorrected visual acuity will be scored for distance, intermediate and near vision:
  * logMAR 0.0 or better = 5
  * logMar 0.1 = 4
  * logMar 0.2 = 3
  * logMar 0.3 = 2
  * logMAR worse than 0.3 = 1 Scores for the individual distances will be added to a total score.
Reading speed and acuity, and preferred reading distance (Salzburg reading desk) | 2-4 Months, & 5-8 Months
  Sites at which the Salzburg Reading Desk is available will examine reading speed and acuity at 40 cm and 66 cm at the two postoperative visits. The following parameters will be documented: words per minute (WPM), characters per minute (CPM), words missed (reading speed recalculated when missed words are selected), LogMAR reading acuity, average reading distance, average reading time.
Postoperative use of spectacles (near, intermediate, distance) | 2-4 Months, & 5-8 Months
  The surgeon asks: "How often do you need glasses for near/intermediate/distance vision?". The answers are classified into 0%, 25%, 50%, 75% and 100% of the total time.
Photic phenomena | 2-4 Months, & 5-8 Months
  The McAlinden Quality of Vision (QoV) questionnaire will be used to assess the size and intensity of halo and glare
Defocus curve | 2-4 Months, & 5-8 Months
  Best-corrected distance defocus curve testing from +1.0 D to -4.0 D shall be performed. The image shall be defocused in -0.5 D increments with spherical minus lenses and a visual acuity measurement is obtained at each defocus increment.
Patient satisfaction | 2-4 Months, & 5-8 Months
  The McAlinden Quality of Vision (QoV) questionnaire will be used to assess patient satisfaction. Patients are asked two closed answered questions, with Yes or No being the answer. 'Would you decide to have multifocal IOLs again?' and ' Would you recommend the same lens to your relatives and friends?'
Surgeon's assessment | 2-4 Months, & 5-8 Months
  The surgeon completes a short questionnaire on the handling and performance of the lens. The ease of implantation, achievement of the target refraction, satisfaction with the patient's vision and general satisfaction are recorded.
Optimization of IOL-constants | 2-4 Months, & 5-8 Months
  For this purpose, the corneal radii, the axial length, the measured anterior chamber depth and the implanted IOL power are recorded during biometry to determine the correct IOL power. Postoperatively, the subjective refraction achieved is documented as spherical equivalent and forwarded to Prof. Dr. Achim Langenbucher, Medical Faculty of Saarland University, Experimental Ophthalmology, for evaluation with the IOL-Con software

CONTACTS AND LOCATIONS:
Overall Officials: Florian Kretz, Principal Investigator — Augentagesklinik Rheine
Locations (4):
- Hellerup Øjenklinik, Hellerup, Denmark
- Germany (2):
  - Goethe University, Frankfurt
  - Augentagesklinik Rheine, Rheine
- Cathedral Eye Clinic, Belfast, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moore J, Ostergaard J, Kretz F. Visual performance and patient preference with bilateral implantation of an extended depth of focus or combined implantation of an extended depth of focus/trifocal intraocular lens. Int Ophthalmol. 2024 Feb 14;44(1):80. doi: 10.1007/s10792-024-03030-y. PMID 38356027